CLINICAL TRIAL: NCT07198074
Title: A Randomized Phase III Trial of Carboplatin, Paclitaxel, Pembrolizumab Versus Carboplatin, Paclitaxel, Bevacizumab Versus Carboplatin, Paclitaxel, Pembrolizumab, Bevacizumab in the Treatment of pMMR, TP53 Mutated Advanced or Recurrent Endometrial Cancer
Brief Title: Testing the Addition of an Antiangiogenic Drug (Bevacizumab) to Chemotherapy (Carboplatin and Paclitaxel) Combined With Immunotherapy (Pembrolizumab) for pMMR, TP53 Mutated Endometrial Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-06974; NCI-2025-06974 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY035 (Other: NRG Oncology); NRG-GY035 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-09-27; First posted 2025-09-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Advanced Endometrial Carcinoma; Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Carboplatin; Magnetic Resonance Spectroscopy; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (paclitaxel, carboplatin, pembrolizumab) (Active Comparator): Patients receive paclitaxel IV over 3 hours, carboplatin IV and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for up to an additional 14 cycles. Additionally, patients undergo urine and blood sample collection and CT or MRI throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab
- Arm 2 (paclitaxel, carboplatin, bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours, carboplatin IV, and bevacizumab IV or anti-VEGF antibody biosimilar on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to an additional 28 doses. Additionally, patients undergo urine and blood sample collection and CT or MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel
- Arm 3 (paclitaxel, carboplatin, pembrolizumab, bevacizumab) (Experimental): Patients receive paclitaxel IV over 3 hours, carboplatin IV, pembrolizumab IV over 30 minutes, and bevacizumab IV or anti-VEGF antibody biosimilar on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance pembrolizumab IV over 30 minutes every 6 weeks for up to an additional 14 cycles and bevacizumab IV every 3 weeks for up to an additional 28 doses. Additionally, patients undergo urine and blood sample collection and CT or MRI throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Paclitaxel; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm 2 (paclitaxel, carboplatin, bevacizumab); Arm 3 (paclitaxel, carboplatin, pembrolizumab, bevacizumab)
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475
  Arms: Arm 1 (paclitaxel, carboplatin, pembrolizumab); Arm 3 (paclitaxel, carboplatin, pembrolizumab, bevacizumab)

SUMMARY:
This phase III trial compares the effect of bevacizumab in combination with carboplatin, paclitaxel and pembrolizumab to the usual treatments of carboplatin and paclitaxel with or without pembrolizumab in treating patients with stage III, IVA or IVB mismatch repair protein proficient (pMMR) and TP53 mutated endometrial cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has come back after a period of improvement (recurrent). Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Carboplatin is in a class of medications known as platinum-containing compounds. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Paclitaxel is in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Adding bevacizumab to the combination of carboplatin, paclitaxel and pembrolizumab may be more effective than the usual treatment combinations of carboplatin and paclitaxel with or without pembrolizumab in treating patients with advanced or recurrent pMMR and TP53 mutated endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that bevacizumab, an anti-VEGF antibody therapy, (or an anti-VEGF antibody biosimilar) in combination with carboplatin, paclitaxel, and pembrolizumab is superior to carboplatin, paclitaxel, and pembrolizumab (the control arm) or carboplatin, paclitaxel, and bevacizumab in prolonging progression-free survival (PFS) in patients with pMMR, TP53 mutated advanced stage (III or IV) or recurrent endometrial cancer.

SECONDARY OBJECTIVES:

I. To demonstrate that bevacizumab in combination with carboplatin, paclitaxel, and pembrolizumab is superior to carboplatin, paclitaxel, and pembrolizumab or carboplatin, paclitaxel, and bevacizumab in prolonging overall survival (OS) in patients with pMMR, TP53 mutated advanced stage (III or IV) or recurrent endometrial cancer.

II. To examine the impact of the addition of bevacizumab in combination with carboplatin and paclitaxel or with carboplatin, paclitaxel, and pembrolizumab on PFS and OS based on type of p53 immunohistochemistry (IHC) aberrancy (over expression/cytoplasmic expression versus null [complete absence of staining]) and mutation type.

III. To evaluate toxicity on treatment with bevacizumab when combined with carboplatin, paclitaxel, and/or pembrolizumab as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.)5.0.

IV. To explore the anti-tumor activity in each treatment arm as assessed by objective response rate in the subset of patients with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM 1 (REFERENCE ARM): Patients receive paclitaxel intravenously (IV) over 3 hours, carboplatin IV and pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for up to an additional14 cycles. Additionally, patients undergo urine and blood sample collection and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study.

ARM 2 (EXPERIMENTAL TRIPLET ARM): Patients receive paclitaxel IV over 3 hours, carboplatin IV, and bevacizumab IV or anti-VEGF antibody biosimilar on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to an additional 28 doses. Additionally, patients undergo urine and blood sample collection and CT or MRI throughout the study.

ARM 3 (EXPERIMENTAL QUADRUPLET ARM): Patients receive paclitaxel IV over 3 hours, carboplatin IV, pembrolizumab IV over 30 minutes, and bevacizumab IV or anti-VEGF antibody biosimilar on day 1 of each cycle. Cycles repeat every 3 weeks for up to 6-10 cycles in the absence of disease progression or unacceptable toxicity. Starting 3 weeks after last combination phase cycle, patients may continue to receive maintenance pembrolizumab IV over 30 minutes every 6 weeks for up to an additional 14 cycles and bevacizumab IV every 3 weeks for up to an additional 28 doses. Additionally, patients undergo urine and blood sample collection and CT or MRI throughout the study.

After completion of study treatment, patients are followed every 3 months for 2 years then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of disease:

  * Stage III and stage IVA endometrial cancers (with measurable disease),
  * Stage IVB endometrial cancer (with or without measurable disease), or
  * Recurrent endometrial cancer (with or without measurable disease)
* In patients with measurable disease, lesions will be defined and monitored by RECIST 1.1. Measurable disease (RECIST 1.1) is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT or MRI. Lymph nodes must be ≥ 15 mm in short axis when measured by CT or MRI
* Histologic confirmation of the original primary tumor is required (submission of pathology report[s] is required). Patients with the following histologic types are eligible: endometrioid, serous, dedifferentiated/undifferentiated, clear cell, mixed epithelial, carcinosarcoma, adenocarcinoma not otherwise specified (N.O.S.)
* Patients must have:

  * Tumoral mismatch repair proficient (pMMR) disease as assessed by immunohistochemistry (IHC) AND
  * P53 IHC with aberrant staining pattern (aberrant p53 expression is consistent with mutant TP53). TP53 mutation by next-generation sequencing will also be accepted
* A pathology report demonstrating results of institutional MMR IHC and p53 IHC and/or TP53 by next-generation sequencing
* Patients may have received:

  * NO prior chemotherapy for treatment of endometrial cancer OR
  * Prior adjuvant chemotherapy (e.g., paclitaxel/carboplatin alone or as a component of concurrent chemotherapy and radiation therapy [with or without cisplatin]) provided adjuvant chemotherapy was completed ≥ 12 months prior to registration
* Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para-aortic radiation therapy, intravaginal brachytherapy, and/or palliative radiation therapy. All radiation therapy must be completed at least 4 weeks prior to registration. For patients with recent radiation, they must have RECIST-evaluable disease outside of the radiation field and have recovered their marrow function
* Patients may have received prior hormonal (endocrine) therapy. All hormonal (endocrine) therapy must have been completed at least 1 week prior to registration
* NO prior pembrolizumab (or other anti-PD1, anti-PDL1 or anti-CTLA4 therapy) or bevacizumab (or other antiangiogenic therapy)
* Interval or cytoreductive surgery, after start of treatment on this trial, and prior to documentation of disease progression, is NOT permitted
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of disease progression. Patients with brain metastases must have follow up imaging demonstrating no evidence of disease progression and that the disease is stable off of steroids
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Not pregnant and not nursing
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8 g/dl
* Creatinine clearance (CrCl) of ≥ 30 mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level ≤ 3 x institutional ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x institutional ULN
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* No active infection requiring parenteral antibiotics
* No current evidence of intra-abdominal abscess, abdominal/pelvic fistula (not diverted), gastrointestinal perforation, gastrointestinal (GI) obstruction, and/or need for drainage nasogastric or gastrostomy tube
* No clinically significant bleeding within 28 days prior to registration
* No uncontrolled hypertension, defined as systolic ≥ 160 mm Hg or diastolic ≥ 100 mm Hg
* No major surgery within 28 days of initiation of bevacizumab
* No active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including corticosteroids. This includes, but is not limited to, patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome because of the risk of recurrence or exacerbation of disease

  * Patients with vitiligo, endocrine deficiencies including type I diabetes mellitus, thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible
  * Topical or inhaled steroids are allowed
  * Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), and anti-thyroid antibodies should be evaluated with the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* No history of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* No history of stem cell or solid organ transplant
* No history of allergic reaction to the study agent(s) or compounds of similar chemical or biologic composition to the study agent(s) (or any of its excipients)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years
  Will be defined using Response Evaluation Criteria in Solid Tumors version (v) 1.1. Will be tested using one-sided log-rank tests with α-levels stratified by factors used in the randomization. Patients will be grouped by their randomized treatment assignment for intention-to-treat (ITT) analyses, supported by patients in ITT population. Treatment hazard ratios and their 95% confidence intervals will be estimated using a Cox proportional hazards models specified with a main effect for the randomized treatment assignment and stratified using the stratification factors applied at randomization.

SECONDARY OUTCOMES:
Overall survival (OS) | From study entry to time of death from any cause, assessed up to 5 years
  Will be assessed with proportional hazards modeling stratified for stratification factors at baseline. Hazard ratios and corresponding 2-sided 95% confidence intervals will be estimated for treatment (with Arm 1 as the reference arm).
Prognostic and predictive associations of type of TP53 mutation status with PFS | Up to 5 years
  Will be assessed with proportional hazards modeling stratified for stratification factors at baseline and adjusted by randomized treatment arm assignment. Hazard ratios and corresponding 2-sided 95% confidence intervals will be estimated for TP53 status as well as treatment hazard ratios (with Arm 1 as the reference arm) within TP53 subgroups.
Prognostic and predictive associations of type of TP53 mutation status with OS | Up to 5 years
  Will be assessed with proportional hazards modeling stratified for stratification factors at baseline and adjusted by randomized treatment arm assignment. Hazard ratios and corresponding 2-sided 95% confidence intervals will be estimated for TP53 status as well as treatment hazard ratios (with Arm 1 as the reference arm) within TP53 subgroups.
Incidence of adverse events (AEs) in treatment with bevacizumab when combined with carboplatin, paclitaxel, and pembrolizumab | Up to 90 days after last dose of study treatment
  The nature, frequency, and degree of toxicity will be tabulated at the system organ class and AE-specific term levels using Common Terminology Criteria for Adverse Events v 5.0. Each patient will be represented according to maximum grade observed for each term. Tabulations will show the number and percentage of patients by maximum grade, within the treatment group received, regardless of the randomized treatment assignment. No specific hypothesis test is pre-specified.
Objective response rate | Within 12 months of initiating therapy
  Will be defined as the binomial proportion of evaluable patients with a best overall response of complete response or partial response. Will be supported by their 2-sided, 95% Wilson-Score confidence intervals. The relative odds of response in each experimental group (vs the reference group) will be estimated using a multivariable logistic regression model specified with main effects for the treatment groups and stratified by the stratification factors reported at baseline.

OTHER OUTCOMES:
PFS | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years
  Will estimate the PFS treatment effect and the corresponding 95% confidence intervals by sex.
PFS | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years
  Will estimate the PFS treatment effect and the corresponding 95% confidence intervals by race.
PFS | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years
  Will estimate the PFS treatment effect and the corresponding 95% confidence intervals by ethnicity.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda N Fader, Principal Investigator — NRG Oncology
Locations (26):
- United States (26):
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital Springfield, Springfield, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Community Medical Center, Missoula, Montana
  - ProMedica Flower Hospital, Sylvania, Ohio
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm